CLINICAL TRIAL: NCT04751201
Title: Meditation and Cancer: Effectiveness of the MAEva Program on Symptoms and Quality of Life. Pilot Feasibility Study. (MAEva Pilot Study)
Brief Title: Meditation and Cancer, Pilot Feasibility Study (MAEva Pilot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A03205-34
Record Dates: First submitted 2021-02-04; First posted 2021-02-12 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; Prostate Cancer
Keywords: Mindfulness; Quality of life; Cancer; Open and circular program; Meditation
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receiving mindfulness open and circular program (Experimental)
  Interventions: Behavioral: Mindfulness open and circular program

INTERVENTIONS:
Behavioral: Mindfulness open and circular program — At the end of the first and the last cycle, as well as 3 weeks after the last cycle, the patient will be invited to answer different questionnaires evaluating his or her quality of life (HADS, QLQC30, FA12). This is why the observation period is 3 months (3 cycles of 3 weeks + 3 weeks).
  Similarly, some of the patients included in the study will be asked to complete a semi-structured interview at the end of the MAEva programme.
  Patients and nursing staff participating in the study will be asked to complete a satisfaction questionnaire

SUMMARY:
MAEVA, which stands for Meditation, Acceptance and Commitment towards Values, is an open and circular program, made up of 3 themed sessions, following a weekly rhythm. It is proposed here to study this program over a period of 3 months, which will give participants the opportunity to complete up to three complete cycles.

This program is based on the practice of and the processes of acceptance and commitment therapy. These approaches, used for several years, have proven their effectiveness in the management of stress, chronic anxiety, insomnia, chronic pain, distress in the face of chronic disease, as well as in the prevention of depressive relapses and management of impulsivity.

Unlike conventional 8-week meditation programs, the MAEva program allows patients to enter the study at any stage of the disease (within, outside the exclusion criteria) and from any session and to participate according to their possibilities.

The patient can participate in a weekly session of the program for 3 cycles. During the sessions, it will be proposed to train meditative practices and 3 different themes will be addressed (one theme per session): Meditation, Acceptance and Commitment to values.

.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient with non-metastatic prostate or breast cancer
* Newly diagnosed patients or those undergoing treatment
* Patient able and willing to follow all study procedures in accordance with the protocol.
* Patient having understood, signed and dated the consent form.
* Patient affiliated to the social security system
* Patient able to remain in a sitting position during the 2-hour session

Exclusion Criteria:

* Impossibility to undergo the medical follow-up of the trial for geographical, social or psychological reasons.
* Presence of an acute psychiatric disorder: depression in acute phase, unstabilised bipolar disorder, psychotic disorders (delusions, hallucinations), etc.
* Presence of recurrent uncontrolled panic attacks (notably linked to hypochondriac concerns)
* Presence of latent or patent post-traumatic stress disorder
* Lack of motivation to meditate
* Insufficient attentional resources to meditate: major problems with attention, memory or reasoning
* Patient with metastatic cancer.
* Presence of cognitive and neurocognitive disorders and deficits
* Presence of deafness
* Membership in a meditation programme prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility and acceptability of the MAEva programme to patients in a specialised care facility | 3 months
  Patient participation rate and number of sessions performed per patient

SECONDARY OUTCOMES:
Improved patient well-being | 3 months
  Hospital Anxiety et Depression Scale (HADS) and Quality of Life Questionnaire C30 (QLQC30) and QLQ -FA12 (EORTC Cancer Related Fatigue)
Measure patient satisfaction | 3 months
  Satisfaction questionnaire [1: unsatisfied - 10 very satisfied]
Measure care staff satisfaction | 3 months
  Satisfaction questionnaire [1: unsatisfied - 10 very satisfied]

CONTACTS AND LOCATIONS:
Overall Officials: François Bourgognon, PhD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Bourgognon F, Bechet D, Huin-Schohn C, Strelow A, Demarche L, Guillou M, Adam V, Fall E, Omorou AY. A mixed method feasibility and acceptability study of a flexible intervention based on acceptance and commitment therapy for patients with cancer. Front Psychol. 2024 Jul 3;15:1409308. doi: 10.3389/fpsyg.2024.1409308. eCollection 2024. PMID 39021646